CLINICAL TRIAL: NCT05987956
Title: Explore the Relationship Between Single Nucleotide Polymorphisms and Alectinib Response and Toxicity in Patients With Non-Small Cell Lung Cancer.
Brief Title: Pharmacogenomics IND EXEMPT SNP Clinical Study - Alectinib and Single Nucleotide Polymorphisms
Acronym: Drugs-SNPs
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair (Industry)
Collaborators: UnitedHealthcare (Other)
Responsible Party: Sponsor-Investigator, Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, M.D., Ph.D., Sponsor-Investigator, Medical Director, Medical Monitor, Safety Officer, IRB Chair, Medicine Invention Design, Inc
Organization: Medicine Invention Design, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IND 168453; FWA00015357 (Registry Identifier: HHS, Human Protections Administrator); NPI - 1831468511 (Registry Identifier: HHS, Health Care Provider Individual); NPI - 1023387701 (Registry Identifier: HHS, Health Care Provider Organization); IRB00009424 (Registry Identifier: HHS, IRB); IORG0007849 (Registry Identifier: HHS, IORG); IND 168453 (Registry Identifier: FDA, IND)
Record Dates: First submitted 2023-07-29; First posted 2023-08-14 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: ALK; EGFR; NSCLC; SNP; Pharmacogenomics; Gene; Genetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: * The usual approach group (NDC...01)
  * The study approach group (NDC...86)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: No-placebo and random and double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alectinib - Usual (Experimental): * Usual ALECENSA - Alectinib
  * Chemotherapy (NDC...01)
  * Usual ALECENSA - alectinib hydrochloride capsule 600 mg orally twice daily
  * Usual Approach Group (NDC...01)
  * ALECENSA - alectinib hydrochloride capsule -- 600 mg orally twice daily
  Interventions: Drug: Alectinib - Usual
- Alectinib - Study (Experimental): * Study ALECENSA - Alectinib
  * Chemotherapy (NDC...86)
  * Study ALECENSA - alectinib hydrochloride capsule 600 mg orally twice daily
  * Study Approach Group (NDC...86)
  * ALECENSA - alectinib hydrochloride capsule -- 600 mg orally twice daily
  Interventions: Drug: Alectinib - Study

INTERVENTIONS:
Drug: Alectinib - Usual — Usual Alectinib Chemotherapy (NDC...01)
  - ALECENSA - alectinib hydrochloride capsule -- 600 mg orally twice daily
  Other Names: Usual ALECENSA - alectinib hydrochloride capsule 600 mg orally twice daily
  Arms: Alectinib - Usual
Drug: Alectinib - Study — Study Alectinib Chemotherapy (NDC...86)
  - ALECENSA - alectinib hydrochloride capsule -- 600 mg orally twice daily
  Other Names: Study ALECENSA - alectinib hydrochloride capsule 600 mg orally twice daily
  Arms: Alectinib - Study

SUMMARY:
Explore the relationship between drug target ALK gene single nucleotide polymorphisms and ALECENSA - Alectinib therapeutic-effects in patients with non-small cell lung cancer, based on Oxford precisely sequencing drug targets' genes.

Explore the relationship between drug target CYP4503A4 gene single nucleotide polymorphisms and ALECENSA - Alectinib side-effects in patients with non-small cell lung cancer, based on Oxford precisely sequencing drug targets' genes.

DETAILED DESCRIPTION:
The usual approach group, after biopsy diagnosis, 300 double blind random group separated NSCLC patients currently used the Chemotherapy on ALECENSA - alectinib hydrochloride capsule 600 mg orally twice daily, it will try to look for the relationship between the Alectinib therapeutic efficacy and the ALK SNP Genotyping, and the relationship between the Alectinib therapeutic safety and the CYP4503A SNP Genotyping, based on Oxford precisely sequencing drug targets' genes.

The study approach group, after biopsy diagnosis, 300 double blind random group separated NSCLC patients currently used the Chemotherapy on ALECENSA - alectinib hydrochloride capsule 600 mg orally twice daily, it will try to look for the relationship between the Alectinib therapeutic efficacy and the ALK SNP Genotyping, and the relationship between the Alectinib therapeutic safety and the CYP4503A4 SNP Genotyping, based on Oxford precisely sequencing drug targets' genes.

1. Detect drug target whole gene precision sequence of everyone patient for all 600 recruited double blind NSCLC patients.
2. Mutually compare everyone patient drug target whole gene precision sequence for a total of 600 recruited double blind NSCLC patients.
3. Calculate drug target gene SNPs in all 600 recruited double blind NSCLC patients.
4. Correlate everyone patient drug target gene SNP to everyone patient drug efficacy.
5. Correlate everyone patient drug target gene SNP to everyone patient drug safety.
6. Mutually compare the usual approach group SNPs (300 double blind random group separated NSCLC patients) with the study approach group SNPs (300 double blind random group separated NSCLC patients).
7. Confirm the relationship between drug target gene SNPs and drug efficacy.
8. Confirm the relationship between drug target gene SNPs and drug safety.

ELIGIBILITY:
* Select 600 Non-Small Cell Lung Cancer Patients who are suitable for blood-drawing.
* Dosage Duration at least 90 days
* The usual approach group - Recruit 300 double blind random group separated NSCLC patients currently used the Chemotherapy NDC...01 on ALECENSA - alectinib hydrochloride capsule 600 mg orally twice daily, film coated after biopsy diagnosis, like as the usual approach group.
* The study approach group - Recruit 300 double blind random group separated NSCLC patients currently used the Chemotherapy NDC...86 on ALECENSA - alectinib hydrochloride capsule 600 mg orally twice daily, film coated after biopsy diagnosis, like as the study approach group.

Inclusion Criteria:

* 1. Clinical diagnosis of Non-Small Cell Lung Cancer (NSCLC)
* 2. Clinical biopsy diagnosis of NSCLC
* 3. Suitable for enough blood-drawing
* 4. Random and double blind
* 5. Measurable disease
* 6. Adequate organ functions
* 7. Adequate performance status
* 8. Age 22 years old and over
* 9. Sign an informed consent form
* 10. Receive blood-drawing

Exclusion Criteria:

* 1. Pneumonectomy
* 2. Treatment with other anti-cancer therapies and cannot be stopped currently
* 3. Pregnancy
* 4. Breast-feeding
* 5. The patients with other serious intercurrent illness or infectious diseases
* 6. Have more than one different kind of cancer at the same time
* 7. Serious Allergy to Drugs
* 8. Serious Bleed Tendency
* 9. Serious Risks or Serious Adverse Events of the drug product
* 10. The prohibition of drug products
* 11. Have no therapeutic effects
* 12. Follow up to the most current label

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-11-08 (Estimated); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Measure and Report Alectinib Drug Targets' SNP Genotypes which are effectiveness-associated, and which are risk-associated. | Up to 12 weeks
  * Recruit 300 double blind random group separated NSCLC patients currently using the Chemotherapy NDC...01 on ALECENSA - alectinib 600 mg orally twice daily, after biopsy diagnosis, to be the usual approach group.
  * Recruit 300 double blind random group separated NSCLC patients currently using the Chemotherapy NDC...86 on ALECENSA - alectinib 600 mg orally twice daily, after biopsy diagnosis, to be the study approach group.
  * Measure above every NSCLC patient-specific Alectinib drug target (ALK) SNP genotype in his or her WBC cell whole genome DNA with Oxford precisely sequencing.
  * Report every NSCLC patient-specific ALK SNP genotype in whole genome DNA sequence.
  * Measure above every NSCLC patient-specific Alectinib drug target (CYP4503A4) SNP genotype in his or her WBC cell whole genome DNA with Oxford precisely sequencing.
  * Report every NSCLC patient-specific CYP4503A4 SNP genotype in whole genome DNA sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Han Xu, MD/PhD/FAPCR, Principal Investigator — Medicine Invention Design, Inc. - IORG0007849; Han Xu, MD/PhD/FAPCR, Study Director — Medicine Invention Design, Inc. - IORG0007849; Han Xu, MD/PhD/FAPCR, Study Chair — Medicine Invention Design, Inc. - IORG0007849
Locations (1):
- Medicine Invention Design, Inc. - IORG0007849, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FWA < 00015357 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search
- See also: IRB < 00009424 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search
- See also: IORG < 0007849 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search

DOCUMENTS (3):
  • Study Protocol (2023-12-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT05987956/Prot_013.pdf
  • Statistical Analysis Plan (2023-12-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT05987956/SAP_014.pdf
  • Informed Consent Form (2023-12-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT05987956/ICF_015.pdf